CLINICAL TRIAL: NCT03092336
Title: Effects of Different Protocols of Physical Training on Levels of Muscle Strength and Functional Capacity on Patients With Peripheral Artery Disease: a Randomized Clinical Trial
Brief Title: Effects of Different Protocols of Physical Training on Levels of Muscle Strength and Functional Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-0566
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease, training
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Electric Stimulation; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation (Experimental): The training with electrostimulation will be performed with the following intensity:
  Medium frequency current: 2.500Hz Modulation frequency: up to 50Hz Time on / off: 1: 2 Average session time 10 to 15 min Being applied in the same muscle groups that will be trained in the group that will perform strength training.
  Interventions: Other: Electrical Stimulation
- Strength training (Experimental): There will be 10 exercises: upper limbs: Supine with dumbbells; High pulley pull; Alternating thread with dumbbells; Triceps dumbbell test; Lower limbs: knee extensor, squatting with body weight, plantar flexion, knee flexion and plantar dorsiflexion. The session time will be from 45 minutes to one hour 2 times weekly totaling at the end of the 12 weeks, 24 strength training sessions.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Electrical Stimulation — electrical stimulation training
  Arms: Electrical Stimulation
Other: Strength training — strength training group
  Arms: Strength training

SUMMARY:
Introduction: the peripheral obstructive arterial disease is an condition that affects around 15% of the world population interfering in muscle strength, life quality and functional capacity of patients.

DETAILED DESCRIPTION:
Study aim: to assess three methods of physical training (strength training, aerobic training and electrical stimulation training) in muscle strength, functional capacity and life quality of patients with peripheral obstructive arterial disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAD and IC.
* Age from 40 to 80 years.
* Stage I and II of Fontaine.
* Symptoms of Intermittent Claudication for at least 3 months with resting brachial index ≤ 0.90 in 1 or 2 legs

Exclusion Criteria:

* Critical ischemia in one of the lower limbs.
* Moderate or severe ulcers in one of the lower limbs. Orthopedic problems that prevent exercise or evaluation.
* Participation in other studies with rehabilitation.
* Decreased arterial hypertension.
* Decompensated Diabetes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2011-05 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
cardiopulmonary exercise test | 13 months
  assess functional capacity

SECONDARY OUTCOMES:
WHOQOL Questionnaire | 13 months
  asses quality of life
Brachial ultrasonography | 13 months
  endothelial function
Analog scale of pain | 13 months
  assess pain intensity
Repetition maximum strength test (1RM) | 13 months
  assess Muscle strengh

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Santos, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia LA. Epidemiology and pathophysiology of lower extremity peripheral arterial disease. J Endovasc Ther. 2006 Feb;13 Suppl 2:II3-9. doi: 10.1177/15266028060130S204. PMID 16472007
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Gardner AW, Montgomery PS, Afaq A. Exercise performance in patients with peripheral arterial disease who have different types of exertional leg pain. J Vasc Surg. 2007 Jul;46(1):79-86. doi: 10.1016/j.jvs.2007.02.037. Epub 2007 May 30. PMID 17540534
- [Background] Chi YW, Jaff MR. Optimal risk factor modification and medical management of the patient with peripheral arterial disease. Catheter Cardiovasc Interv. 2008 Mar 1;71(4):475-89. doi: 10.1002/ccd.21401. PMID 18307227
- [Background] Makdisse M, Pereira Ada C, Brasil Dde P, Borges JL, Machado-Coelho GL, Krieger JE, Nascimento Neto RM, Chagas AC; Hearts of Brazil Study and Peripheral Arterial Disease Committee of the Brazilian Society of Cardiology/Funcor. Prevalence and risk factors associated with peripheral arterial disease in the Hearts of Brazil Project. Arq Bras Cardiol. 2008 Dec;91(6):370-82. doi: 10.1590/s0066-782x2008001800008. PMID 19142364
- [Background] Kullo IJ, Bailey KR, Kardia SL, Mosley TH Jr, Boerwinkle E, Turner ST. Ethnic differences in peripheral arterial disease in the NHLBI Genetic Epidemiology Network of Arteriopathy (GENOA) study. Vasc Med. 2003 Nov;8(4):237-42. doi: 10.1191/1358863x03vm511oa. PMID 15125483
- [Background] Selvin E, Erlinger TP. Prevalence of and risk factors for peripheral arterial disease in the United States: results from the National Health and Nutrition Examination Survey, 1999-2000. Circulation. 2004 Aug 10;110(6):738-43. doi: 10.1161/01.CIR.0000137913.26087.F0. Epub 2004 Jul 19. PMID 15262830
- [Background] Garg PK, Tian L, Criqui MH, Liu K, Ferrucci L, Guralnik JM, Tan J, McDermott MM. Physical activity during daily life and mortality in patients with peripheral arterial disease. Circulation. 2006 Jul 18;114(3):242-8. doi: 10.1161/CIRCULATIONAHA.105.605246. Epub 2006 Jul 3. PMID 16818814
- [Background] Askew CD, Green S, Walker PJ, Kerr GK, Green AA, Williams AD, Febbraio MA. Skeletal muscle phenotype is associated with exercise tolerance in patients with peripheral arterial disease. J Vasc Surg. 2005 May;41(5):802-7. doi: 10.1016/j.jvs.2005.01.037. PMID 15886664
- [Background] Bendermacher BL, Willigendael EM, Teijink JA, Prins MH. Supervised exercise therapy versus non-supervised exercise therapy for intermittent claudication. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005263. doi: 10.1002/14651858.CD005263.pub2. PMID 16625633
- [Background] Murphy TP, Hirsch AT, Ricotta JJ, Cutlip DE, Mohler E, Regensteiner JG, Comerota AJ, Cohen DJ; CLEVER Steering Committee. The Claudication: Exercise Vs. Endoluminal Revascularization (CLEVER) study: rationale and methods. J Vasc Surg. 2008 Jun;47(6):1356-63. doi: 10.1016/j.jvs.2007.12.048. Epub 2008 Apr 25. PMID 18440181
- [Background] Andreozzi GM, Leone A, Laudani R, Deinite G, Martini R. Acute impairment of the endothelial function by maximal treadmill exercise in patients with intermittent claudication, and its improvement after supervised physical training. Int Angiol. 2007 Mar;26(1):12-7. PMID 17353883
- [Background] European Stroke Organisation; Tendera M, Aboyans V, Bartelink ML, Baumgartner I, Clement D, Collet JP, Cremonesi A, De Carlo M, Erbel R, Fowkes FG, Heras M, Kownator S, Minar E, Ostergren J, Poldermans D, Riambau V, Roffi M, Rother J, Sievert H, van Sambeek M, Zeller T; ESC Committee for Practice Guidelines. ESC Guidelines on the diagnosis and treatment of peripheral artery diseases: Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteries: the Task Force on the Diagnosis and Treatment of Peripheral Artery Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2011 Nov;32(22):2851-906. doi: 10.1093/eurheartj/ehr211. Epub 2011 Aug 26. No abstract available. PMID 21873417
- [Background] Treesak C, Kasemsup V, Treat-Jacobson D, Nyman JA, Hirsch AT. Cost-effectiveness of exercise training to improve claudication symptoms in patients with peripheral arterial disease. Vasc Med. 2004 Nov;9(4):279-85. doi: 10.1191/1358863x04vm570oa. PMID 15678620
- [Background] Ambrosetti M, Salerno M, Boni S, Daniele G, Tramarin R, Pedretti RF. Economic evaluation of a short-course intensive rehabilitation program in patients with intermittent claudication. Int Angiol. 2004 Jun;23(2):108-13. PMID 15507886
- [Background] Hiatt WR, Wolfel EE, Meier RH, Regensteiner JG. Superiority of treadmill walking exercise versus strength training for patients with peripheral arterial disease. Implications for the mechanism of the training response. Circulation. 1994 Oct;90(4):1866-74. doi: 10.1161/01.cir.90.4.1866. PMID 7923674
- [Background] Parr BM, Noakes TD, Derman EW. Peripheral arterial disease and intermittent claudication: efficacy of short-term upper body strength training, dynamic exercise training, and advice to exercise at home. S Afr Med J. 2009 Nov;99(11):800-4. PMID 20218480
- [Background] McGuigan MR, Bronks R, Newton RU, Sharman MJ, Graham JC, Cody DV, Kraemer WJ. Resistance training in patients with peripheral arterial disease: effects on myosin isoforms, fiber type distribution, and capillary supply to skeletal muscle. J Gerontol A Biol Sci Med Sci. 2001 Jul;56(7):B302-10. doi: 10.1093/gerona/56.7.b302. PMID 11445595
- [Background] Anderson SI, Whatling P, Hudlicka O, Gosling P, Simms M, Brown MD. Chronic transcutaneous electrical stimulation of calf muscles improves functional capacity without inducing systemic inflammation in claudicants. Eur J Vasc Endovasc Surg. 2004 Feb;27(2):201-9. doi: 10.1016/j.ejvs.2003.10.003. PMID 14718904
- [Background] Kelsall CJ, Brown MD, Kent J, Kloehn M, Hudlicka O. Arteriolar endothelial dysfunction is restored in ischaemic muscles by chronic electrical stimulation. J Vasc Res. 2004 May-Jun;41(3):241-51. doi: 10.1159/000078301. Epub 2004 Apr 30. PMID 15118363
- [Background] Presern-Strukelj M, Poredos P. The influence of electrostimulation on the circulation of the remaining leg in patients with one-sided amputation. Angiology. 2002 May-Jun;53(3):329-35. doi: 10.1177/000331970205300311. PMID 12025921
- [Background] Zwierska I, Walker RD, Choksy SA, Male JS, Pockley AG, Saxton JM. Upper- vs lower-limb aerobic exercise rehabilitation in patients with symptomatic peripheral arterial disease: a randomized controlled trial. J Vasc Surg. 2005 Dec;42(6):1122-30. doi: 10.1016/j.jvs.2005.08.021. PMID 16376202
- [Background] Ratliff DA, Puttick M, Libertiny G, Hicks RC, Earby LE, Richards T. Supervised exercise training for intermittent claudication: lasting benefit at three years. Eur J Vasc Endovasc Surg. 2007 Sep;34(3):322-6. doi: 10.1016/j.ejvs.2007.04.014. Epub 2007 Jun 22. PMID 17587612
- [Background] Campeau L, Enjalbert M, Lesperance J, Bourassa MG, Kwiterovich P Jr, Wacholder S, Sniderman A. The relation of risk factors to the development of atherosclerosis in saphenous-vein bypass grafts and the progression of disease in the native circulation. A study 10 years after aortocoronary bypass surgery. N Engl J Med. 1984 Nov 22;311(21):1329-32. doi: 10.1056/NEJM198411223112101. PMID 6333635
- [Background] Watson NL, Sutton-Tyrrell K, Youk AO, Boudreau RM, Mackey RH, Simonsick EM, Rosano C, Hardy SE, Windham BG, Harris TB, Najjar SS, Lakatta EG, Atkinson HH, Johnson KC, Bauer DC, Newman AB; Health ABC Study. Arterial stiffness and gait speed in older adults with and without peripheral arterial disease. Am J Hypertens. 2011 Jan;24(1):90-5. doi: 10.1038/ajh.2010.193. Epub 2010 Sep 9. PMID 20940711
- [Background] Monahan KD, Tanaka H, Dinenno FA, Seals DR. Central arterial compliance is associated with age- and habitual exercise-related differences in cardiovagal baroreflex sensitivity. Circulation. 2001 Oct 2;104(14):1627-32. doi: 10.1161/hc3901.096670. PMID 11581140
- [Background] Parmenter BJ, Raymond J, Dinnen P, Singh MA. A systematic review of randomized controlled trials: Walking versus alternative exercise prescription as treatment for intermittent claudication. Atherosclerosis. 2011 Sep;218(1):1-12. doi: 10.1016/j.atherosclerosis.2011.04.024. Epub 2011 May 5. PMID 21601857
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Rabkin SW, Chan SH, Sweeney C. Ankle-brachial index as an indicator of arterial stiffness in patients without peripheral artery disease. Angiology. 2012 Feb;63(2):150-4. doi: 10.1177/0003319711410307. Epub 2011 Jun 15. PMID 21676966
- [Background] Parmenter BJ, Raymond J, Fiatarone Singh MA. The effect of exercise on fitness and performance-based tests of function in intermittent claudication: a systematic review. Sports Med. 2013 Jun;43(6):513-24. doi: 10.1007/s40279-013-0038-9. PMID 23539309
- [Background] Kruidenier LM, Viechtbauer W, Nicolai SP, Buller H, Prins MH, Teijink JA. Treatment for intermittent claudication and the effects on walking distance and quality of life. Vascular. 2012 Feb;20(1):20-35. doi: 10.1258/vasc.2011.ra0048. Epub 2012 Jan 23. PMID 22271802
- [Background] McDermott MM, Ades P, Guralnik JM, Dyer A, Ferrucci L, Liu K, Nelson M, Lloyd-Jones D, Van Horn L, Garside D, Kibbe M, Domanchuk K, Stein JH, Liao Y, Tao H, Green D, Pearce WH, Schneider JR, McPherson D, Laing ST, McCarthy WJ, Shroff A, Criqui MH. Treadmill exercise and resistance training in patients with peripheral arterial disease with and without intermittent claudication: a randomized controlled trial. JAMA. 2009 Jan 14;301(2):165-74. doi: 10.1001/jama.2008.962. PMID 19141764
- [Background] Adams J, Ogola G, Stafford P, Koutras P, Hartman J. High-intensity interval training for intermittent claudication in a vascular rehabilitation program. J Vasc Nurs. 2006 Jun;24(2):46-9. doi: 10.1016/j.jvn.2006.03.002. PMID 16737929
- [Background] Lee HL, Mehta T, Ray B, Heng MS, McCollum PT, Chetter IC. A non-randomised controlled trial of the clinical and cost effectiveness of a Supervised Exercise Programme for claudication. Eur J Vasc Endovasc Surg. 2007 Feb;33(2):202-7. doi: 10.1016/j.ejvs.2006.08.005. Epub 2006 Dec 4. PMID 17142065
- [Background] Wang J, Zhou S, Bronks R, Graham J, Myers S. Effects of supervised treadmill walking training on calf muscle capillarization in patients with intermittent claudication. Angiology. 2009 Feb-Mar;60(1):36-41. doi: 10.1177/0003319708317337. Epub 2008 May 27. PMID 18505746
- [Background] Roberts AJ, Roberts EB, Sykes K, De Cossart L, Edwards P, Cotterrell D. Physiological and functional impact of an unsupervised but supported exercise programme for claudicants. Eur J Vasc Endovasc Surg. 2008 Sep;36(3):319-24. doi: 10.1016/j.ejvs.2008.04.008. Epub 2008 Jun 10. PMID 18547828
- [Background] Gardner AW, Killewich LA, Montgomery PS, Katzel LI. Response to exercise rehabilitation in smoking and nonsmoking patients with intermittent claudication. J Vasc Surg. 2004 Mar;39(3):531-8. doi: 10.1016/j.jvs.2003.08.037. PMID 14981444
- [Background] Atkins LM, Gardner AW. The relationship between lower extremity functional strength and severity of peripheral arterial disease. Angiology. 2004 Jul-Aug;55(4):347-55. doi: 10.1177/000331970405500401. PMID 15258680
- [Background] McDermott MM, Guralnik JM, Albay M, Bandinelli S, Miniati B, Ferrucci L. Impairments of muscles and nerves associated with peripheral arterial disease and their relationship with lower extremity functioning: the InCHIANTI Study. J Am Geriatr Soc. 2004 Mar;52(3):405-10. doi: 10.1111/j.1532-5415.2004.52113.x. PMID 14962156
- [Background] Scott-Okafor HR, Silver KK, Parker J, Almy-Albert T, Gardner AW. Lower extremity strength deficits in peripheral arterial occlusive disease patients with intermittent claudication. Angiology. 2001 Jan;52(1):7-14. doi: 10.1177/000331970105200102. PMID 11205935
- [Background] Regensteiner JG, Wolfel EE, Brass EP, Carry MR, Ringel SP, Hargarten ME, Stamm ER, Hiatt WR. Chronic changes in skeletal muscle histology and function in peripheral arterial disease. Circulation. 1993 Feb;87(2):413-21. doi: 10.1161/01.cir.87.2.413. PMID 8425290
- [Background] Parmenter BJ, Raymond J, Dinnen PJ, Lusby RJ, Fiatarone Singh MA. Preliminary evidence that low ankle-brachial index is associated with reduced bilateral hip extensor strength and functional mobility in peripheral arterial disease. J Vasc Surg. 2013 Apr;57(4):963-973.e1. doi: 10.1016/j.jvs.2012.08.103. Epub 2012 Dec 14. PMID 23246081
- [Background] Smart NA, Dieberg G, Giallauria F. Functional electrical stimulation for chronic heart failure: a meta-analysis. Int J Cardiol. 2013 Jul 15;167(1):80-6. doi: 10.1016/j.ijcard.2011.12.019. Epub 2012 Jan 10. PMID 22236510
- [Background] Vivodtzev I, Debigare R, Gagnon P, Mainguy V, Saey D, Dube A, Pare ME, Belanger M, Maltais F. Functional and muscular effects of neuromuscular electrical stimulation in patients with severe COPD: a randomized clinical trial. Chest. 2012 Mar;141(3):716-725. doi: 10.1378/chest.11-0839. Epub 2011 Nov 23. PMID 22116795
- [Background] Black CD, Elder CP, Gorgey A, Dudley GA. High specific torque is related to lengthening contraction-induced skeletal muscle injury. J Appl Physiol (1985). 2008 Mar;104(3):639-47. doi: 10.1152/japplphysiol.00322.2007. Epub 2007 Dec 13. PMID 18079265
- [Background] Hortobagyi T, Dempsey L, Fraser D, Zheng D, Hamilton G, Lambert J, Dohm L. Changes in muscle strength, muscle fibre size and myofibrillar gene expression after immobilization and retraining in humans. J Physiol. 2000 Apr 1;524 Pt 1(Pt 1):293-304. doi: 10.1111/j.1469-7793.2000.00293.x. PMID 10747199
- [Background] Hamilton MT, Booth FW. Skeletal muscle adaptation to exercise: a century of progress. J Appl Physiol (1985). 2000 Jan;88(1):327-31. doi: 10.1152/jappl.2000.88.1.327. PMID 10642397
- [Background] Green HJ, Pette D. Early metabolic adaptations of rabbit fast-twitch muscle to chronic low-frequency stimulation. Eur J Appl Physiol Occup Physiol. 1997;75(5):418-24. doi: 10.1007/s004210050182. PMID 9189729
- [Background] Skorjanc D, Jaschinski F, Heine G, Pette D. Sequential increases in capillarization and mitochondrial enzymes in low-frequency-stimulated rabbit muscle. Am J Physiol. 1998 Mar;274(3):C810-8. doi: 10.1152/ajpcell.1998.274.3.C810. PMID 9530113
- [Background] Hudlicka O, Milkiewicz M, Cotter MA, Brown MD. Hypoxia and expression of VEGF-A protein in relation to capillary growth in electrically stimulated rat and rabbit skeletal muscles. Exp Physiol. 2002 May;87(3):373-81. doi: 10.1113/eph8702285. PMID 12089605
- [Background] Milkiewicz M, Hudlicka O, Verhaeg J, Egginton S, Brown MD. Differential expression of Flk-1 and Flt-1 in rat skeletal muscle in response to chronic ischaemia: favourable effect of muscle activity. Clin Sci (Lond). 2003 Oct;105(4):473-82. doi: 10.1042/CS20030035. PMID 12780346
- [Background] Egginton S, Hudlicka O. Selective long-term electrical stimulation of fast glycolytic fibres increases capillary supply but not oxidative enzyme activity in rat skeletal muscles. Exp Physiol. 2000 Sep;85(5):567-73. PMID 11038408